CLINICAL TRIAL: NCT01482065
Title: The Sleep, Liver Evaluation and Effective Pressure Study (SLEEP)
Brief Title: The Sleep, Liver Evaluation and Effective Pressure Study
Acronym: SLEEP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: ResMed Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00048965; 111481 (Other Grant/Funding Number: ResMed Foundation)
Record Dates: First submitted 2011-11-15; First posted 2011-11-30 (Estimated); Results first posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-11

CONDITIONS: Non Alcoholic Fatty Liver Disease; Obstructive Sleep Apnea
Keywords: Non Alcoholic Fatty Liver Disease; NAFLD; Continuous Positive Airway Pressure; CPAP; CPAP Therapy; Apnea Hypopnea Index; Non alcoholic steatohepatitis; NASH; OSA; Obstructive Sleep Apnea; AHI
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CPAP (Experimental): Patients with moderate to severe apnea will be randomized to CPAP or deferred CPAP. Those in the CPAP group will be sent home with an autoset CPAP device, which they will be instructed to utilize for 4 months. The CPAP device will be set in the "auto mode" so that it will automatically adjust the pressure at night to eliminate upper airway obstruction during sleep.
  Criteria for OSA severity are specifically designed to target patients with nocturnal hypoxemia, which is hypothesized to contribute to NAFLD progression. According to the guidelines of the American Academy of Sleep Medicine, apnea will be defined as cessation of airflow for ≥ 10 sec. and hypopnea will be defined as decreased airflow for ≥ 10 sec. leading to oxyhemoglobin desaturation ≥ 4%. Mild, moderate and severe OSA will be diagnosed by an Apnea-Hypopnea Index (AHI) of 5-14.9, 15-29.9, and ≥ 30 events/hr, respectively.
  Interventions: Device: CPAP (ResMed S9 autoset CPAP)

INTERVENTIONS:
Device: CPAP (ResMed S9 autoset CPAP) — A ResMed S9 autoset CPAP device will be utilized throughout the study. Throughout the study intervention period, subjects (for AHI> 15) will be instructed to utilize their CPAP and adherence will be monitored using an automatic meter that is built into the CPAP device.
  Other Names: ResMed S9 autoset CPAP

SUMMARY:
This research is being done to examine: 1) how common obstructive sleep apnea (OSA) is in patients with non-alcoholic fatty liver disease (NAFLD), 2) whether the severity of OSA is related to the severity of NAFLD, and 3) whether treatment of OSA with continuous positive airway pressure (CPAP) improved NAFLD progression.

OSA is a condition caused by repetitive collapse of throat tissue during sleep that leads to falls in oxygen level and sleep disruption. OSA can be caused by obesity, and especially by fat found in the neck and belly.

NAFLD is a common disease linked to obesity. NAFLD is part of a disease spectrum, which can progress from steatosis (fatty liver) to nonalcoholic steatohepatitis (NASH), a progressive fibrotic disease, in which cirrhosis and liver-related death can occur. Recent evidence in patients with obstructive sleep apnea (OSA) indicates that OSA is associated with NASH. How common OSA is in patients with biopsy-confirmed NAFLD and the effect of OSA treatment with CPAP on NASH is unknown.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is a common disease with a well-established link to obesity and is increasingly prevalent with the concurrent rise in obesity. NAFLD constitutes a disease spectrum from steatosis to cirrhosis and is associated with significant morbidity and mortality. The pathogenesis of NAFLD, especially disease progression, is not well understood. Obesity and insulin resistance play a role as 'a first hit' leading to liver steatosis, but the mechanisms for a 'second hit' triggering progression to steatohepatitis are not known. Based on our Preliminary Data, we propose a novel hypothesis that chronic intermittent hypoxia (CIH) in patients with obstructive sleep apnea (OSA) constitutes a 'second hit' causing progression of NAFLD from steatosis to nonalcoholic steatohepatitis (NASH), a progressive fibrotic disease, in which cirrhosis and liver-related death occur in up to 20% and 12% patients, respectively.

Obstructive sleep apnea (OSA) is characterized by recurrent collapse of the upper airway during sleep, leading to CIH. OSA is a common disease, present in 2% of women and 4% of men in the general US population, but with an increased prevalence of 30-60% in obese populations. Furthermore, CIH has been associated with multiple metabolic complications of OSA independent of obesity, including insulin resistance, dyslipidemia, and atherosclerosis. Previous work in rodent models has demonstrated that intermittent hypoxia (IH) increases: (1) insulin resistance; (2) hepatic steatosis; (3) hepatic levels of Sterol regulatory element-binding protein-1 (SREBP-1) and Stearoyl-CoA desaturase (SCD-1); and (4) hepatic oxidative stress and inflammation Thus, CIH in OSA may contribute to hepatic steatosis, and convert hepatic steatosis to steatohepatitis. To address this hypothesis, we will establish the impact of OSA on NASH in a susceptible cohort of obese human subjects in whom definitive intraoperative liver biopsy will be available to diagnose and stage NAFLD.

Recent evidence in patients with obstructive sleep apnea (OSA) indicates that OSA is associated with NASH. Nevertheless, the prevalence of OSA in patients with biopsy-confirmed NAFLD is unknown and the effect of OSA treatment with CPAP on NASH has never been studied. Our main hypothesis is that the severity of nocturnal intermittent hypoxemia of obstructive sleep apnea (OSA) will be associated with the severity of NAFLD. We will examine NAFLD severity in patients with and without obstructive sleep apnea and examine the effect of CPAP on NAFLD progression in patients with obstructive sleep apnea.

The overall goal is to determine whether OSA is associated with NAFLD and whether CPAP mitigates NAFLD progression. Our primary hypothesis is that the severity of nocturnal intermittent hypoxemia of obstructive sleep apnea (OSA) will be associated with the severity of NAFLD.

* In Specific Aim #1, we will examine NAFLD severity in patients with and without obstructive sleep apnea. We hypothesize that the severity of NAFLD and the presence of NASH will be associated with the presence and severity of OSA.
* In Specific Aim #2, we will examine the effect of CPAP on NAFLD progression in patients with obstructive sleep apnea. We hypothesize that CPAP will decrease markers of hepatic inflammation (serum aminotransferases) in patients with NAFLD, who have moderate or severe OSA. To address this hypothesis, we will enroll patients from the Johns Hopkins Medical Institution (JHMI) Hepatology clinic with the diagnosis of NAFLD, who have elevated serum aminotransferases, NAFLD on liver biopsy, and moderate to severe OSA. The effect of CPAP on markers of liver inflammation and serum aminotransferases will be determined, and related to CPAP adherence.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21
* Diagnosis of NAFLD and BMI ≥ 30 or obesity with BMI > 35 and < 400lbs
* No other cause of liver disease other than NAFLD (as assessed by patient and physician surveys detailed below, blood work and magnetic resonance imaging(MRI))

Exclusion Criteria:

Both patients and doctors will be asked to identify potential exclusionary conditions including:

1. Patients with sickle cell anemia, hemoglobinopathies and other hemolytic anemias
2. Known clinical hypersensitivity or a history of asthma or allergic respiratory disorders
3. Advanced renal failure (currently requiring dialysis or with a Glomerular Filtration rate < 30cc/min)
4. Pregnancy
5. History of CPAP treatment for OSA
6. Recent weight loss (6 months) ≥ 10%
7. Current alcohol use > 20 g/day in women and > 30 g/day in men, or prior use for ≥ 3 consecutive months during the previous 5 years as assessed with the Lifetime Drinking History Questionnaire Viral hepatitis A, B and C
8. Autoimmune hepatitis
9. Hemochromatosis
10. Wilson's disease
11. Alpha-1-antitrypsin deficiency
12. Primary sclerosing cholangitis
13. Cirrhosis of any etiology
14. History of HIV infection and/or HAART therapy
15. Evidence of drug-induced liver injury
16. Use of systemic steroids for > 10 days during prior 6 months
17. Unstable cardiovascular disease (decompensated chronic heart failure (CHF), myocardial infarction or revascularization procedures, unstable arrhythmias)
18. Uncontrolled hypertension with BP > 190/110
19. Daytime hypoxemia with oxygen saturation (SaO2)<90%
20. Supplemental oxygen use
21. Presence of any contraindication to MR examinations (see MRI Safety Screening Sheet)
22. History of Metal in the Skull/Eyes
23. Unable to have an MRI Scan
24. Severe daytime hypersomnolence as defined by an Epworth Sleepiness Score of greater than 10.
25. Severe sleep apnea as characterized by an apnea-hypopnea index of greater than 80 episodes/hour or an average low SaO2 during sleep disordered breathing episodes below 80%.
26. Work in transportation industry as a driver or pilot.
27. Patients with a diagnosis of sleep apnea on active treatment.

Exclusions based on etiology of hepatitis will be assessed by querying both the hepatology list and patient about the above mentioned disorders (#7-15) and through testing for viral hepatitis A, B, C, ferritin, antinuclear antibody (ANA), antineutrophil cytoplasmic antibody (ANCA), anti-mitochondrial antibody, anti-smooth muscle antibody and ceruloplasmin.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-11; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan R Schwartz, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 212 subjects screened; 166 subjects were excluded. 40 were included. 39 started in the protocol. 8 patients dropped out. Liver MRI completed in 27 subjects. 12 patients were excluded after liver MRI; 14 subjects had sleep studies. 5 patients did not proceed to the CPAP trial. 9 patients were randomized.
Groups:
- Deferred CPAP: Patients with moderate to severe apnea will be randomized to CPAP or deferred CPAP. Those in the deferred CPAP group will sign a consent to agree to defer CPAP use for 4 months to complete the study.
  Criteria for Obstructive Sleep Apnea (OSA) severity are specifically designed to target patients with nocturnal hypoxemia, which is hypothesized to contribute to NAFLD progression. According to the guidelines of the American Academy of Sleep Medicine, apnea will be defined as cessation of airflow for ≥ 10 sec. and hypopnea will be defined as decreased airflow for ≥ 10 sec. leading to oxyhemoglobin desaturation ≥ 4%. Mild, moderate and severe OSA will be diagnosed by an AHI of 5-14.9, 15-29.9, and ≥ 30 events/hr, respectively.
  CPAP (ResMed S9 autoset CPAP): A ResMed S9 autoset CPAP device will be utilized throughout the study.
- CPAP: Patients with moderate to severe apnea will be randomized to CPAP or deferred CPAP. Those in the CPAP group will be sent home with an autoset CPAP device, which they will be instructed to utilize for 4 months. The CPAP device will be set in the "auto mode" so that it will automatically adjust the pressure at night to eliminate upper airway obstruction during sleep.
  Criteria for OSA severity are specifically designed to target patients with nocturnal hypoxemia, which is hypothesized to contribute to NAFLD progression. According to the guidelines of the American Academy of Sleep Medicine, apnea will be defined as cessation of airflow for ≥ 10 sec. and hypopnea will be defined as decreased airflow for ≥ 10 sec. leading to oxyhemoglobin desaturation ≥ 4%. Mild, moderate and severe OSA will be diagnosed by an AHI of 5-14.9, 15-29.9, and ≥ 30 events/hr, respectively.
Period: Overall Study
Arm/Group | Deferred CPAP | CPAP
Started | 4 | 5
Completed | 4 | 4
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Deferred CPAP: Patients with moderate to severe apnea will be randomized to CPAP or deferred CPAP. Those in the deferred CPAP group will sign a consent to agree to defer CPAP use for 4 months to complete the study.
  Criteria for OSA severity are specifically designed to target patients with nocturnal hypoxemia, which is hypothesized to contribute to NAFLD progression. According to the guidelines of the American Academy of Sleep Medicine, apnea will be defined as cessation of airflow for ≥ 10 sec. and hypopnea will be defined as decreased airflow for ≥ 10 sec. leading to oxyhemoglobin desaturation ≥ 4%. Mild, moderate and severe OSA will be diagnosed by an AHI of 5-14.9, 15-29.9, and ≥ 30 events/hr, respectively.
  CPAP (ResMed S9 autoset CPAP): A ResMed S9 autoset CPAP device will be utilized throughout the study.
- Total: Total of all reporting groups
Arm/Group | Deferred CPAP | CPAP | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (3.74) | 42.8 (16.63) | 49.56 (14.73)
Gender [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Cross Sectional Analysis of NAFLD Versus Sleep Apnea Severity Indices (AHI)
Description: Cross-sectional analysis will be performed in NAFLD study participants from the Johns Hopkins (JH) Hepatology Clinic to examine the relationship between findings on liver biopsy and sleep apnea severity indices. The main predictor variable will be presence/severity of OSA and nocturnal oxyhemoglobin desaturation (assessed by T90%, time w/ oxyhemoglobin desaturation < 90%; Delta SaO2 between baseline and minimal oxyhemoglobin saturation, and standard deviation of nocturnal SaO2). Our primary outcome will be NAFLD activity score on biopsy.
Time Frame: 6 months
Population: We were unable to obtain liver biopsy on most of our participants due to limited clinical indications.
Arm/Group | Deferred CPAP | CPAP
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Liver Values
Description: Serum Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) activity.
Time Frame: 6 Months
Population: Withdrawal by subject in CPAP group.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Deferred CPAP | CPAP
Number analyzed (Participants) | 4 | 5
U/L
  ALT Baseline | 37.25 (20.66) | 53.8 (27.26)
  ALT 6 Months: number analyzed (Participants) | 4 | 4
  ALT 6 Months | 29 (7.84) | 40.5 (10.36)
  AST Baseline | 26.75 (9.44) | 32.6 (19.77)
  AST 6 Months: number analyzed (Participants) | 4 | 4
  AST 6 Months | 23.5 (7.83) | 29.75 (21.29)

3. Secondary Outcome: Analysis of Variance (ANOVA) in CPAP Versus No-CPAP Therapy on NAFLD
Description: we will test our hypothesis that CPAP therapy improves NAFLD. The main independent variables will be CPAP vs. deferred-CPAP therapy. In a subanalysis, responses in the CPAP treatment group will be compared based on compliance. Compliance with CPAP is defined as using it on > 70% of the days, at least 4 h per night. Our primary outcome will be serum activity of ALT and AST. We will use ANOVA to examine changes in ALT and AST depending on CPAP therapy group and compliance. Secondary outcomes will include the degree of hepatic steatosis and fibrosis, as assessed by MRI.
Time Frame: 6 months
Population: We were unable to achieve enrollment goals due to limited clinical indications. Thereby not obtaining enough participant data to do an Analysis of Variance (ANOVA).
Arm/Group | Deferred CPAP | CPAP
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: MRI Indices
Time Frame: 6 Months
Population: We were not able to obtain MRI data from 2 people within the CPAP group at 6 months. One withdrew from study and the other a clear scan could not be obtained.
Measure: Mean (Standard Deviation); unit: percentage of fat in liver
Arm/Group | Deferred CPAP | CPAP
Number analyzed (Participants) | 4 | 5
percentage of fat in liver
  MRI Baseline | 10.57 (6.33) | 15.406 (3.77)
  MRI 6 Months: number analyzed (Participants) | 4 | 3
  MRI 6 Months | 8.69 (4.82) | 18.76 (11.72)

ADVERSE EVENTS:
Arm/Group | Deferred CPAP | CPAP
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No